CLINICAL TRIAL: NCT01236352
Title: A Phase 1/2 Multiple Ascending Dose Study to Evaluate the Safety, Efficacy, Pharmacokinetics and Pharmacodynamics of BMS-911543 in Subjects With Myelofibrosis
Brief Title: Multiple Ascending Dose of BMS-911543
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to portfolio/business decisions by the sponsor
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA215-001
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Cancer
Keywords: Advanced Cancer, Various, NOS
MeSH Terms: conditions — Neoplasms; Pyloric Stenosis, Hypertrophic | interventions — N,N-dicyclopropyl-4-((1,5-dimethyl-1H-pyrazol-3-yl)amino)-6-ethyl-1-methyl-1,6-dihydroimidazo(4,5-d)pyrrolo(2,3b)pyridine-7-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (12):
- Phase 1 (Cohort 1): BMS-911543 (5 mg) (Experimental): BMS-911543 5 mg capsule by mouth twice daily for 12 months or greater depending on response
  Interventions: Drug: BMS-911543
- Phase 1 (Cohort 2): BMS-911543 (10 mg) (Experimental): BMS-911543 10 mg capsule by mouth twice daily for 12 months or greater depending on response
  Interventions: Drug: BMS-911543
- Phase 1 (Cohort 3): BMS-911543 (20 mg) (Experimental): BMS-911543 20 mg capsule by mouth twice daily for 12 months or greater depending on response
  Interventions: Drug: BMS-911543
- Phase 1 (Cohort 4): BMS-911543 (40 mg) (Experimental): BMS-911543 40 mg capsule by mouth twice daily for 12 months or greater depending on response
  Interventions: Drug: BMS-911543
- Phase 1 (Cohort 5): BMS-911543 (80 mg) (Experimental): BMS-911543 80 mg capsule by mouth twice daily for 12 months or greater depending on response
  Interventions: Drug: BMS-911543
- Phase 1 (Cohort 6): BMS-911543 (120 mg) (Experimental): BMS-911543 120 mg capsule by mouth twice daily for 12 months or greater depending on response
  Interventions: Drug: BMS-911543
- Phase 1 (Cohort 7): BMS-911543 (160 mg) (Experimental): BMS-911543 160 mg capsule by mouth twice daily for 12 months or greater depending on response
  Interventions: Drug: BMS-911543
- Phase 1 (Cohort 8): BMS-911543 (200 mg) (Experimental): BMS-911543 200 mg capsule by mouth twice daily for 12 months or greater depending on response
  Interventions: Drug: BMS-911543
- Phase 1 (Cohort 9): BMS-911543 (240 mg) (Experimental): BMS-911543 240 mg capsule by mouth twice daily for 12 months or greater depending on response
  Interventions: Drug: BMS-911543
- Phase 1 (Cohort 10): BMS-911543 (320 mg) (Experimental): BMS-911543 320 mg capsule by mouth twice daily for 12 months or greater depending on response
  Interventions: Drug: BMS-911543
- Phase 2 (Cohort 11): BMS-911543 (120 mg) (Experimental): BMS-911543 120 mg capsule by mouth twice daily for 12 months or greater depending on response
  Interventions: Drug: BMS-911543
- Phase 2 (Cohort 12): BMS-911543 (200 mg) (Experimental): BMS-911543 200 mg capsule by mouth twice daily for 12 months or greater depending on response
  Interventions: Drug: BMS-911543

INTERVENTIONS:
Drug: BMS-911543
  Other Names: JAK2 Inhibitor

SUMMARY:
The purpose of this first in human study is to determine if BMS-911543 is safe and tolerable in subjects with symptomatic intermediate-1, intermediate-2 or high risk myelofibrosis to permit clinical testing at the Maximum Tolerated Dose or at a Clinically Active Dose, and to determine if BMS-911543 will demonstrate efficacy in symptomatic myelofibrosis.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Men and Women at least 18 years old
* A diagnosis of symptomatic, primary or secondary Myelofibrosis (MF) [World Health Organization (WHO) 2008 criteria] with intermediate-1, intermediate-2 or high risk disease as assessed using the Dynamic International Prognostic Scoring System international prognostic scoring system
* Last therapeutic or diagnostic treatment at least 28 days prior
* Any toxicity from prior therapies must have resolved to Grade ≤1
* Adequate Liver and Kidney Function
* Serum amylase and lipase within normal institutional range
* Platelet count ≥50,000 cell mm³
* Absolute neutrophil count (ANC) ≥1,000 cells/mm3
* Hemoglobin ≥8.0 g/dL

Exclusion Criteria:

* Primary central nervous system tumors
* Subjects with currently active malignancy (other than MF) or with a prior history of malignancy with the exception of: (i) adequately treated basal cell carcinoma of the skin, (ii) curatively treated in situ carcinoma of the cervix, (iii) other malignancy that has undergone potentially curative therapy with no evidence of disease recurrence ≥3 years
* Any condition requiring chronic use of moderate/high dose steroids except inhalation or oral steroids for mild pulmonary disease
* Splenic irradiation ≤3 months prior to treatment with study drug
* Positive blood screen for hepatitis C antibody, hepatitis B surface antigen or Human Immunodeficiency Virus-1 (HIV-1), or HIV-2 antibodies
* Abnormalities in serum electrolytes
* Significant cardiovascular disease
* Current or recent gastrointestinal disease
* Previous history of pancreatitis and/or significant risk factors for pancreatitis as judged by the treating physician
* Evidence of uncontrolled active infection or active graft vs. host disease
* Inability to tolerate oral medication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2011-04-07 (Actual); Primary Completion 2015-11-19 (Actual); Study Completion 2015-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - The Mount Sinai School Of Medicine, New York, New York
  - The University Of Texas Md Anderson Cancer Center, Houston, Texas
- Australia (2):
  - Local Institution, East Melbourne, Victoria
  - Local Institution, Melbourne, Victoria

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 98 participants were enrolled and 84 participants were treated. 14 participants did not enter treatment period (13 no longer met study criteria and 1 due to other reasons). 42 entered Phase 1 and 42 entered Phase 2
Groups:
- 5 mg Phase I: BMS-911543 5 mg capsule by mouth twice daily
- 10 mg Phase I: BMS-911543 10 mg capsule by mouth twice daily
- 20 mg Phase I: BMS-911543 20 mg capsule by mouth twice daily
- 40 mg Phase I: BMS-911543 40 mg capsule by mouth twice daily
- 80 mg Phase I: BMS-911543 80 mg capsule by mouth twice daily
- 120 mg Phase I; 120 mg Phase II: BMS-911543 120 mg capsule by mouth twice daily
- 160 mg Phase I: BMS-911543 160 mg capsule by mouth twice daily
- 200 mg Phase I: BMS-911543 2000 mg capsule by mouth twice daily
- 240 mg Phase I: BMS-911543 240 mg capsule by mouth twice daily
- 200 mg Phase II: BMS-911543 200 mg capsule by mouth twice daily
Period: Overall Study
Arm/Group | 5 mg Phase I | 10 mg Phase I | 20 mg Phase I | 40 mg Phase I | 80 mg Phase I | 120 mg Phase I | 160 mg Phase I | 200 mg Phase I | 240 mg Phase I | 120 mg Phase II | 200 mg Phase II
Started | 4 | 4 | 4 | 4 | 4 | 4 | 8 | 7 | 3 | 22 | 20
Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 4 | 4 | 3 | 4 | 4 | 8 | 7 | 3 | 22 | 20
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 4 | 1
Not completed — Study drug toxicity | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 2
Not completed — Disease progression | 1 | 2 | 1 | 2 | 2 | 2 | 1 | 3 | 2 | 2 | 2
Not completed — Poor/Non-compliance | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Maximum clinical benefit | 1 | 1 | 1 | 0 | 2 | 0 | 3 | 1 | 1 | 4 | 2
Not completed — Subject request to discontinue treatment | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 4
Not completed — Subject to receive drug via EAP | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 0
Not completed — Patient moving to allogeneic transplant | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Relapse of Splenomegaly and symptoms | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of response to drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Patient transferred to IST | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 6

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 mg Phase I | 10 mg Phase I | 20 mg Phase I | 40 mg Phase I | 80 mg Phase I | 120 mg Phase I | 160 mg Phase I | 200 mg Phase I | 240 mg Phase I | 120 mg Phase II | 200 mg Phase II | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 8 | 7 | 3 | 22 | 20 | 84
Age, Continuous [Mean (Standard Deviation); unit: Years] | 76.8 (4.50) | 56.5 (3.70) | 70.5 (4.80) | 64.0 (7.70) | 69.8 (9.54) | 63.3 (12.97) | 70.1 (10.79) | 62.3 (6.47) | 63.0 (6.93) | 61.0 (11.09) | 62.5 (11.13) | 64.0 (10.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 2 | 2 | 2 | 4 | 2 | 1 | 7 | 12 | 39
  Male | 1 | 2 | 2 | 2 | 2 | 2 | 4 | 5 | 2 | 15 | 8 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 00 | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 3 | 3 | 3 | 3 | 4 | 7 | 6 | 3 | 16 | 19 | 70
  Unknown or Not Reported | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 5 | 1 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 4 | 4 | 4 | 4 | 4 | 8 | 7 | 3 | 20 | 20 | 82
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Safety assessments were based on a medical review of adverse event reports and the results of vital sign measurements, ECGs, physical examinations, and clinical laboratory tests and were evaluated for all treated participants using National Cancer Institute Common Terminology Criteria for Adverse Events v4.0 (NCI CTCAE v.4.0).
Time Frame: From the date of participant's written consent until 30 days post discontinuation of dosing or participation in the study if the last scheduled visit occured at a later time, assessed up to 4.5 years
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg Phase I | 10 mg Phase I | 20 mg Phase I | 40 mg Phase I | 80 mg Phase I | 120 mg Phase I | 160 mg Phase I | 200 mg Phase I | 240 mg Phase I | 120 mg Phase II | 200 mg Phase II
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 8 | 7 | 3 | 22 | 20
Participants
  No. of deaths | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 1 | 0
  No. of participants with Serious AEs | 3 | 2 | 2 | 1 | 4 | 2 | 6 | 2 | 1 | 9 | 10
  No. of participants discontinued due to AEs | 1 | 1 | 0 | 0 | 1 | 1 | 3 | 0 | 1 | 7 | 5
  Number of participants with AEs | 4 | 4 | 4 | 4 | 4 | 4 | 8 | 7 | 3 | 22 | 20

2. Primary Outcome: Number of Participants With Best Overall Response
Description: Participants were clinically assessed for IWG-(International Working Group consensus criteria for treatment response in myelofibrosis with myeloid metaplasia) defined response at each returning on-treatment visit and the first post-treatment visit. IWG-MRT criteria for best overall response are ordered high to low: CR>PR>CI>SD>PD>R where CR = Complete Remission, PR= Partial Remission, CI = Clinical Improvement, SD = Stable Disease, PD = Progressive Disease and R = Relapse. Best overall response is the best response of the subject during the treatment period or at the first post-treatment visit.
Time Frame: Day 1, at each returning on-treatment visit and the first post-treatment visit
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg Phase I | 10 mg Phase I | 20 mg Phase I | 40 mg Phase I | 80 mg Phase I | 120 mg Phase I | 160 mg Phase I | 200 mg Phase I | 240 mg Phase I | 120 mg Phase II | 200 mg Phase II
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 8 | 7 | 3 | 22 | 20
Participants
  Complete Remission | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Remission | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  Clinical Improvement | 1 | 1 | 1 | 1 | 2 | 0 | 3 | 3 | 1 | 12 | 9
  Stable Disease | 3 | 2 | 3 | 3 | 1 | 4 | 4 | 3 | 2 | 6 | 10
  Progressive Disease | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Relapse | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Changes in (Janus Kinase) JAK/Signal Transducers and Activators of Transcription (STATs) Pathway Activities, Circulating CD34+ Cells and Plasma Cytokine Levels
Description: JAK/STAT pathway activity will be evaluated by: 1) pSTATs levels using immunoassay; 2) expression levels of several JAK/STATs pathway genes. Whole blood will be collected at specific time-points. Due to portfolio/business decisions by the sponsor, the compound is no longer being developed and the study was terminated. Analysis was not completed because the study was terminated. This decision was not based on any safety concerns associated with BMS-911543.
Time Frame: Up to 6 months
Population: Data for this outcome measure was not collected for any participants because the study was terminated
Arm/Group | 5 mg Phase I | 10 mg Phase I | 20 mg Phase I | 40 mg Phase I | 80 mg Phase I | 120 mg Phase I | 160 mg Phase I | 200 mg Phase I | 240 mg Phase I | 120 mg Phase II | 200 mg Phase II
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of BMS-911543 and it's Metabolite BMS-926796 (Met4)
Description: Pharmacokinetic parameters of BMS-911543 and BMS-926796 (Met4) metabolite, will be derived from plasma concentration versus time. The pharmacokinetic parameters to be assessed include: Cmax Maximum observed plasma concentration
Time Frame: Day -1, Day 1, Day 8, Day 15, Day 21 and Day 28 or off-study
Population: Data for this outcome measure was not collected for any participants because the study was terminated
Arm/Group | 5 mg Phase I | 10 mg Phase I | 20 mg Phase I | 40 mg Phase I | 80 mg Phase I | 120 mg Phase I | 160 mg Phase I | 200 mg Phase I | 240 mg Phase I | 120 mg Phase II | 200 mg Phase II
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Trough Observed (Pre-dose) Plasma Concentration (Cmin) of BMS-911543 and it's Metabolite Met4
Description: Pharmacokinetic parameters of BMS-911543 and BMS-926796 (Met4) metabolite, will be derived from plasma concentration versus time. The pharmacokinetic parameters to be assessed include: Cmin (Trough observed (pre-dose) plasma concentration)
Time Frame: Day -1, Day 1, Day 8, Day 15, Day 21 and Day 28 or off-study
Population: Data for this outcome measure was not collected for any participants because the study was terminated
Arm/Group | 5 mg Phase I | 10 mg Phase I | 20 mg Phase I | 40 mg Phase I | 80 mg Phase I | 120 mg Phase I | 160 mg Phase I | 200 mg Phase I | 240 mg Phase I | 120 mg Phase II | 200 mg Phase II
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Time of Maximum Observed Plasma Concentration (Tmax) of BMS-911543 and it's Metabolite Met4
Description: Pharmacokinetic parameters of BMS-911543 and BMS-926796 (Met4) metabolite, will be derived from plasma concentration versus time. The pharmacokinetic parameters to be assessed include: Tmax = Time of maximum observed plasma concentration (Tmax) of BMS-911543 and it's metabolite Met4
Time Frame: Day -1, Day 1, Day 8, Day 15, Day 21 and Day 28 or off-study
Population: Data for this outcome measure was not collected for any participants because the study was terminated
Arm/Group | 5 mg Phase I | 10 mg Phase I | 20 mg Phase I | 40 mg Phase I | 80 mg Phase I | 120 mg Phase I | 160 mg Phase I | 200 mg Phase I | 240 mg Phase I | 120 mg Phase II | 200 mg Phase II
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinite Time (for Single Dose Period Only) (AUC(INF)) of BMS-911543 and it's Metabolite Met4
Description: Pharmacokinetic parameters of BMS-911543 and BMS-926796 (Met4) metabolite, will be derived from plasma concentration versus time. The pharmacokinetic parameters to be assessed include: AUC(INF) = Area under the plasma concentration-time curve from time zero extrapolated to infinite time (for single dose period only) (AUC(INF)) of BMS-911543 and it's metabolite Met4
Time Frame: Day -1, Day 1, Day 8, Day 15, Day 21 and Day 28 or off-study
Population: Data for this outcome measure was not collected for any participants because the study was terminated
Arm/Group | 5 mg Phase I | 10 mg Phase I | 20 mg Phase I | 40 mg Phase I | 80 mg Phase I | 120 mg Phase I | 160 mg Phase I | 200 mg Phase I | 240 mg Phase I | 120 mg Phase II | 200 mg Phase II
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of Last Quantifiable Plasma Concentration (for Single Dose Period Only) (AUC(0-T)) of BMS-911543 and it's Metabolite Met4
Description: Pharmacokinetic parameters of BMS-911543 and BMS-926796 (Met4) metabolite, will be derived from plasma concentration versus time. The pharmacokinetic parameters to be assessed include: AUC (0-T) = Area under the plasma concentration-time curve from time zero to the time of last quantifiable plasma concentration (for single dose period only) of BMS-911543 and it's metabolite Met4
Time Frame: Day -1, Day 1, Day 8, Day 15, Day 21 and Day 28 or off-study
Population: Data for this outcome measure was not collected for any participants because the study was terminated
Arm/Group | 5 mg Phase I | 10 mg Phase I | 20 mg Phase I | 40 mg Phase I | 80 mg Phase I | 120 mg Phase I | 160 mg Phase I | 200 mg Phase I | 240 mg Phase I | 120 mg Phase II | 200 mg Phase II
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Area Under the Concentration-time Curve in One Dosing Interval (AUC(TAU)) of BMS-911543 and it's Metabolite Met4
Description: Pharmacokinetic parameters of BMS-911543 and BMS-926796 (Met4) metabolite, will be derived from plasma concentration versus time. The pharmacokinetic parameters to be assessed include: AUC (TAU) = Area under the concentration-time curve in one dosing interval of BMS-911543 and it's metabolite Met4
Time Frame: Day -1, Day 1, Day 8, Day 15, Day 21 and Day 28 or off-study
Population: Data for this outcome measure was not collected for any participants because the study was terminated
Arm/Group | 5 mg Phase I | 10 mg Phase I | 20 mg Phase I | 40 mg Phase I | 80 mg Phase I | 120 mg Phase I | 160 mg Phase I | 200 mg Phase I | 240 mg Phase I | 120 mg Phase II | 200 mg Phase II
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: The Terminal-phase Elimination Half-life in Plasma (T-HALF) of BMS-911543 and it's Metabolite Met4
Description: Pharmacokinetic parameters of BMS-911543 and BMS-926796 (Met4) metabolite, will be derived from plasma concentration versus time. The pharmacokinetic parameters to be assessed include: T-HALF = The terminal-phase elimination half-life in plasma of BMS-911543 and it's metabolite Met4
Time Frame: Day -1, Day 1, Day 8, Day 15, Day 21 and Day 28 or off-study
Population: Data for this outcome measure was not collected for any participants because the study was terminated
Arm/Group | 5 mg Phase I | 10 mg Phase I | 20 mg Phase I | 40 mg Phase I | 80 mg Phase I | 120 mg Phase I | 160 mg Phase I | 200 mg Phase I | 240 mg Phase I | 120 mg Phase II | 200 mg Phase II
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Apparent Total Clearance (for Parent Compound Only) (CLT/F) of BMS-911543 and it's Metabolite Met4
Description: Pharmacokinetic parameters of BMS-911543 and BMS-926796 (Met4) metabolite, will be derived from plasma concentration versus time. The pharmacokinetic parameters to be assessed include: CLT/F = Apparent total clearance (for parent compound only) of BMS-911543 and it's metabolite Met4
Time Frame: Day -1, Day 1, Day 8, Day 15, Day 21 and Day 28 or off-study
Population: Data for this outcome measure was not collected for any participants because the study was terminated
Arm/Group | 5 mg Phase I | 10 mg Phase I | 20 mg Phase I | 40 mg Phase I | 80 mg Phase I | 120 mg Phase I | 160 mg Phase I | 200 mg Phase I | 240 mg Phase I | 120 mg Phase II | 200 mg Phase II
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Apparent Volume of Distribution After First Dosing Based on the Terminal Phase (for Parent Compound Only) (Vz/F) of BMS-911543 and it's Metabolite Met4
Description: Pharmacokinetic parameters of BMS-911543 and BMS-926796 (Met4) metabolite, will be derived from plasma concentration versus time. The pharmacokinetic parameters to be assessed include: Vz/F = Apparent volume of distribution after first dosing based on the terminal phase (for parent compound only) of BMS-911543 and it's metabolite Met4
Time Frame: Day -1, Day 1, Day 8, Day 15, Day 21 and Day 28 or off-study
Population: Data for this outcome measure was not collected for any participants because the study was terminated
Arm/Group | 5 mg Phase I | 10 mg Phase I | 20 mg Phase I | 40 mg Phase I | 80 mg Phase I | 120 mg Phase I | 160 mg Phase I | 200 mg Phase I | 240 mg Phase I | 120 mg Phase II | 200 mg Phase II
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Accumulation Index (AI): Ratio of AUC(TAU) on Day 15 to AUC(TAU) After the First Dose of BMS-911543 and it's Metabolite Met4
Description: Pharmacokinetic parameters of BMS-911543 and BMS-926796 (Met4) metabolite, will be derived from plasma concentration versus time. The pharmacokinetic parameters to be assessed include: Accumulation index (AI) = ratio of AUC(TAU) on Day 15 to AUC(TAU) after the first dose of BMS-911543 and it's metabolite Met4
Time Frame: Day -1, Day 1, Day 8, Day 15, Day 21 and Day 28 or off-study
Population: Data for this outcome measure was not collected for any participants because the study was terminated
Arm/Group | 5 mg Phase I | 10 mg Phase I | 20 mg Phase I | 40 mg Phase I | 80 mg Phase I | 120 mg Phase I | 160 mg Phase I | 200 mg Phase I | 240 mg Phase I | 120 mg Phase II | 200 mg Phase II
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Ratio of BMS-926796 AUC(INF) to BMS-911543 AUC(INF) After 1st Dose and BMS-926796 AUC(TAU) to BMS-911543 AUC(TAU) on Day 15 (AUC Ratio)
Description: Pharmacokinetic parameters of BMS-911543 and BMS-926796 (Met4) metabolite, will be derived from plasma concentration versus time. The pharmacokinetic parameters to be assessed include: AUC Ratio = Ratio of BMS-926796 AUC(INF) to BMS-911543 AUC(INF) after 1st dose and BMS-926796 AUC(TAU) to BMS-911543 AUC(TAU) on Day 15
Time Frame: Day -1, Day 1, Day 8, Day 15, Day 21 and Day 28 or off-study
Population: Data for this outcome measure was not collected for any participants because the study was terminated
Arm/Group | 5 mg Phase I | 10 mg Phase I | 20 mg Phase I | 40 mg Phase I | 80 mg Phase I | 120 mg Phase I | 160 mg Phase I | 200 mg Phase I | 240 mg Phase I | 120 mg Phase II | 200 mg Phase II
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the date of subject's written consent until 30 days post discontinuation of dosing or subject's participation in the study if the last scheduled visit occurs at a later time (approximately 4.5 years)
Arm/Group | 5 mg Phase I | 10 mg Phase I | 20 mg Phase I | 40 mg Phase I | 80 mg Phase I | 120 mg Phase I | 160 mg Phase I | 200 mg Phase I | 240 mg Phase I | 120 mg Phase II | 200 mg Phase II
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/4 | 0/4 | 0/4 | 1/4 | 1/4 | 1/8 | 2/7 | 0/3 | 1/22 | 0/20
Serious Adverse Events (participants affected / at risk) | 3/4 | 2/4 | 2/4 | 1/4 | 4/4 | 2/4 | 6/8 | 2/7 | 1/3 | 9/22 | 10/20
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 4/4 | 4/4 | 4/4 | 4/4 | 8/8 | 7/7 | 3/3 | 22/22 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 5 mg Phase I (N=4) | 10 mg Phase I (N=4) | 20 mg Phase I (N=4) | 40 mg Phase I (N=4) | 80 mg Phase I (N=4) | 120 mg Phase I (N=4) | 160 mg Phase I (N=8) | 200 mg Phase I (N=7) | 240 mg Phase I (N=3) | 120 mg Phase II (N=22) | 200 mg Phase II (N=20)
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atypical mycobacterial lymphadenitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroentiritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Listeriosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spleen disorder (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0/0 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Adenosquamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood pressure inadequately controlled (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 5 mg Phase I (N=4) | 10 mg Phase I (N=4) | 20 mg Phase I (N=4) | 40 mg Phase I (N=4) | 80 mg Phase I (N=4) | 120 mg Phase I (N=4) | 160 mg Phase I (N=8) | 200 mg Phase I (N=7) | 240 mg Phase I (N=3) | 120 mg Phase II (N=22) | 200 mg Phase II (N=20)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 3 | 2 | 1 | 4 | 7 | 4 | 2 | 17 | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 2 | 1 | 1 | 4 | 2 | 2 | 3 | 9
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 3 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 3
Spleen disorder (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0
Fatigue (General disorders) | 1 | 3 | 3 | 0 | 2 | 1 | 2 | 5 | 1 | 3 | 6
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 1 | 4 | 4
Oedema (General disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 2 | 2
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 3 | 2
Influenza like illness (General disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 2
Early satiety (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2
Oedema peripheral (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 2 | 2 | 1 | 2 | 2 | 4 | 1 | 6 | 10
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 3 | 2 | 0 | 2 | 1 | 2 | 0 | 7 | 8
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 2 | 0 | 1 | 3 | 1 | 7 | 4
Abdominal Pain (Gastrointestinal disorders) | 2 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 7 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | 1 | 2 | 2 | 4 | 1 | 6 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 3 | 2 | 2 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 4 | 5
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 2 | 10 | 8
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 3 | 6
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 0 | 1 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 0 | 3 | 4
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 1 | 2 | 2
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Lipase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 7
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 3 | 6
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 2
Weight decreased (Investigations) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Amylase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 4 | 1 | 7 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 5 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 3 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0 | 2 | 1 | 2 | 0 | 3 | 3
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 2 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 5 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 1 | 2 | 2 | 0 | 3 | 2 | 1 | 8
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 2
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 2 | 5
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 3
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.